CLINICAL TRIAL: NCT02987920
Title: A Randomized Double-blinded Study to Evaluate Preincisional Dextromethorphan in Patients Undergoing Total Knee Arthroplasty and Its Effect on Postoperative Opioid Use
Brief Title: Dextromethorphan Use in Multimodal Analgesia Regimens for Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The surgeon changed pain control protocol for all patients. Continued enrollment impossible under approved protocol.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Hanna Schittek, Clinical Assistance Professor of Anesthesiology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-16-00739
Record Dates: First submitted 2016-11-30; First posted 2016-12-09 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dextromethorphan; Acetaminophen; Oxycodone; Celecoxib; Pantoprazole; Ketorolac; Ketorolac Tromethamine; Gabapentin; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo - Concentrate (Active Comparator): preoperative oral medications given one time: acetaminophen 1000mg tablet, oxycodone extended release 10mg tablet, celecoxib 400mg tablet, pantoprazole 40mg tablet, and Placebo - Concentrate by mouth.
  postoperative medications given for 2 days: Acetaminophen 1000mg every 6hr, Ketorolac15mg IV q6hrs x4 doses, Oxycodone 5mg po q3hrs prn moderate pain, Oxycodone10mg po q3hrs prn severe pain, Gabapentin100-300mg once at night, Dilaudid 0.2mg IV q2hrs prn severe pain
  Interventions: Drug: Placebo - Concentrate; Drug: Acetaminophen; Drug: Oxycodone; Drug: Celecoxib; Drug: Pantoprazole; Drug: Ketorolac; Drug: Gabapentin; Drug: Hydromorphone
- Dextromethorphan (Experimental): preoperative oral medications given one time: acetaminophen 1000mg tablet, oxycodone extended release 10mg tablet, celecoxib 400mg tablet, pantoprazole 40mg tablet, and Dextromethorphan 60mg tablet
  postoperative medications given for 2 days: Acetaminophen 1000mg every 6hr, Ketorolac15mg IV q6hrs x4 doses, Oxycodone 5mg po q3hrs prn moderate pain, Oxycodone10mg po q3hrs prn severe pain, Gabapentin100-300mg once at night, Dilaudid 0.2mg IV q2hrs prn severe pain, and dextromethorphan 60mg by mouth twice daily
  Interventions: Drug: Dextromethorphan; Drug: Acetaminophen; Drug: Oxycodone; Drug: Celecoxib; Drug: Pantoprazole; Drug: Ketorolac; Drug: Gabapentin; Drug: Hydromorphone

INTERVENTIONS:
Drug: Dextromethorphan — Additional medication to perioperative analgesic regimen in Group B
  Other Names: delsym
  Arms: Dextromethorphan
Drug: Placebo - Concentrate — Additional medication to perioperative analgesic regimen to Group A
  Other Names: placebo, placebos, sugar water
  Arms: Placebo - Concentrate
Drug: Acetaminophen — Multimodal analgesic regimen to Group A and Group B
  Other Names: tylenol
Drug: Oxycodone — Multimodal analgesic regimen to Group A and Group B
  Other Names: oxycodone extended release; oxycontin
Drug: Celecoxib — Multimodal analgesic regimen to Group A and Group B
  Other Names: celebrex
Drug: Pantoprazole — Multimodal analgesic regimen to Group A and Group B
  Other Names: protonix
Drug: Ketorolac — Multimodal analgesic regimen to Group A and Group B
  Other Names: toradol
Drug: Gabapentin — Multimodal analgesic regimen to Group A and Group B
  Other Names: neurontin
Drug: Hydromorphone — Multimodal analgesic regimen to Group A and Group B
  Other Names: dilaudid

SUMMARY:
Total knee arthroplasty (TKA) is one of the most painful orthopedic procedures. After TKA surgery, postoperative pain relief may be achieved using a variety of techniques. Integral to recovery and improved outcomes is early ambulation and mobilization. Achieving adequate postoperative pain control while ensuring the ability to ambulate early can be quite challenging.

Currently, in our country there has been a call to address prescription opioid use and abuse due to a nationwide opioid epidemic. In light of this, improving our multimodal analgesic protocol will serve to decrease reliance of opioid medications for pain control. Multimodal analgesia is effective in decreasing total opioid consumption postoperatively. Dextromethorphan is a low-affinity noncompetitive N-methyl-D-aspartate (NMDA) receptor antagonist. It has a long history of clinical use with an established safety record. Studies have shown that it has a positive effect as an analgesic.

In order to see if dextromethorphan will decrease opioid use, this study will look at two patient groups undergoing total knee arthroplasty with the same preoperative, intraoperative, and postoperative anesthetic plan with the exception of the addition of dextromethorphan to one groups multimodal analgesic regimen. This study is designed as a double-blinded, randomized, prospective cohort trial.

DETAILED DESCRIPTION:
Each subject will receive as part of their standard of care a spinal with sedation for intraoperative anesthesia.

Subjects will be randomly assigned using computer generated allotment. The group designation will be placed in sealed envelopes. The group listed will determine whether or not they will receive dextromethorphan as part of their preoperative preincisional analgesic regimen. Only the pharmacist dispensing the medication will be unblinded. The drug and placebo will then be concealed by the pharmacist and delivered to the patient to ingest in the preoperative area.

Group A: standard preop meds

Group B: standard preop meds + dextromethorphan

The standard preoperative analgesic regimen will include placement of an adductor canal catheter nerve block, acetaminophen 1000mg PO, oxycodone extended release 10mg PO, celecoxib 400mg PO (held if elevated creatinine), and pantoprazole 40mg PO

All blocks will be performed by resident trainees under the supervision of anesthesia regional and acute pain attendings. The continuous adductor canal nerve block will be placed using B-Braun "Contiplex Continuous Peripheral Nerve Block Tray", using 20g catheters.

Intraoperative anesthesia will be performed with spinal injection using local anesthestic only. No opioid will be given intrathecally. Intraoperative sedation will include standard sedation with propofol infusion. Postoperative nausea and vomiting prophylaxis will include ondansetron, propofol infusion, and dexamethasone 0.1mg/kg if not contraindicated. The postoperative recovery room pain protocol will include the following: starting the adductor canal catheter infusion with "On-Q" pump dispensing ropivicaine 0.1% at 4ml/hr, oxycodone 5 10mg po for moderate to severe pain, dilaudid 0.2mg IV q5min up to 2 mg, ketorolac 30mg intravenous (IV) once, and acetaminophen 1000mg intravenous once if greater than 6 hours has elapsed since initial preoperative dose.

Assessments of pain using the VAS pain score will be performed in postanesthesia care unit (PACU) at the time of spinal block cessation by a blinded observer (recovery room nurse), and then subsequently every 4 hours by a registered nurse and documented in the electronic medical record. Initial evaluation for resolution of the spinal blockade will be performed at the 1 hour timepoint in the PACU.

Assessments of opioid administration, will include all medications given and documented in the electronic medical record. The various time points analyzed will include intraoperative, PACU, and daily postoperative morphine equivalents administered to each patient.

Postoperative followup will be done by research personnel blinded to the group distribution. Visual Analog Scale for Pain (VAS Pain) will be performed every 4 hours until discharge.

On postoperative day (POD) #1, all patients will be given the Quality of Recovery (QoR) Questionnaire. This is recovery specific, patient rated questionnaire containing 40 items measuring 5 dimensions. The QoR 40 was specifically designed to measure a patient's health status after surgery and anesthesia, and its completion time generally ranges from 3 to 10 min. The five dimensions measured include: the physical comfort (12 items), emotional state (nine items), physical independence (five items), psychological support (seven items) and pain (seven items). The total score and subscales of the QoR 40 are measured using a five point Likert scale (for positive items: 1 = none of the time, 5 = all of the time; for negative items, the scoring was reversed) and individual scores are then added together, with the minimum score being 40 points and the maximum score being 200 points.

In addition, the study will require home follow up phone calls assessing the occurrence of any possible side effects or complications, pain, and postoperative opioid use. These phone calls will occur at POD#3 after discharge, POD #7, POD #14, and POD#28. Each of these phone assessments will require about 5 minutes of time. Authorized research personnel of the study project will be making the phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age, American Society of Anesthesiologists (ASA) > IIII) who are undergoing only elective primary total knee replacement will be included in the study.

Exclusion Criteria:

* patient refusal to be included in the study, contraindications to regional anesthesia, history of allergy to amide local anesthetics, the presence of a progressive neurological deficit, chronic pain diagnoses, the presence of coagulopathy or infection, or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Total amount of postoperative opioid used in first 48 hours after knee replacement. | 48 hours

SECONDARY OUTCOMES:
VAS pain scores | 28 days

OTHER OUTCOMES:
Total postoperative opioid requirements | Through study completion, an average of 1 year
Presence of postoperative nausea and vomiting | 24 hours
  Will ask patient if they felt nauseated or had any episodes of emesis within the first 24 hours postoperatively. Will obtain yes or no answer to nausea and emesis specifically
Duration of adductor canal catheter | 72 hours
Length of hospital stay | 72 hours
Patient satisfaction questionnaire | 4 weeks
  Patients will be called after discharged from hospital to go through a questionnaire to assess their satisfaction with pain control

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Schittek, MD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No